CLINICAL TRIAL: NCT06507033
Title: Development of the Wearable Arm Volume Measurement Device and Mobile Application (mobiLymphf) in the Prevention and Early Detection of Breast Cancer-related Lymphedema and Evaluation of Their Efficiency
Brief Title: Development of the Wearable Arm Volume Measurement Device and Mobile Application
Acronym: mobiLymphf
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe ARIKAN DÖNMEZ (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor-Investigator, Ayşe ARIKAN DÖNMEZ, Assoc. Prof., Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 223S524
Record Dates: First submitted 2024-06-27; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer Related Lymphedema
Keywords: Breast Cancer; Lymphedema; Wearable Technology; Mobile Application; Nursing
MeSH Terms: conditions — Breast Cancer Lymphedema; Breast Neoplasms; Lymphedema

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): This group will be provided with the mobile application and volume measurement device. The planning for hospital visits will be organised at the same frequency in both groups. All individuals will be followed up for three months. The same measurement tools will be applied to both groups before and after the application.
  Interventions: Device: Mobile application and an arm volume measurement device
- Control Group (No Intervention): This group will receive routine care at the clinic.The planning for hospital visits will be organised at the same frequency in both groups. All individuals will be followed up for three months. The same measurement tools will be applied to both groups before and after the application.

INTERVENTIONS:
Device: Mobile application and an arm volume measurement device — The intervention consists mainly of two steps; (a) development of a mobile application with an arm volume measurement device (b) evaluation of the effectiveness of the products. Five components will be involved in the development of the mobile application. These components are; (I) exercise, (II) education, (III) coping mechanisms, (IV) arm volume measurement/recording and (V) appointment, exercise and measurement reminder panel. Exercise videos will include stretching exercises for the shoulder and arm as recommended in the guidelines
  Arms: Intervention Group

SUMMARY:
With the increase in the incidence of cancer in our country and the world, the number of breast cancer survivors is increasing rapidly due to the development of early diagnosis and treatment methods. One of the main problems in breast cancer survivors is lymphedema. Breast cancer-related lymphedema is a condition that can be treated when detected early, but has a very low success rate when detected in advanced stages. Therefore, the prevention and early detection of breast cancer-associated lymphedema is very important. In this project, it is aimed to prevent breast cancer-related lymphedema with the mobile application to be developed and to detect the volume increase in the arm before clinical findings with an arm volume measurement device that will work with this mobile application. The project consists of two main steps; (a)development of the arm volume measuring device and mobile application (b)evaluation of the effectiveness of the products. Five components will be involved in the development of the mobile application. These components are; (I)exercise, (II)education, (III)coping mechanisms, (IV)arm volume measurement/records, and (V)reminder for exercise, measurement, and follow-ups. Exercise videos will include stretching exercises for the shoulder and arm area as recommended in the guides. The training content will be created in line with the guides and opinions will be taken from an expert panel. In support of coping mechanisms, existing problem areas in people will be determined with a qualitative study. People who have gone through a similar process in the past will be asked about the coping strategies they have developed for these problem areas. Themes obtained from patients who have gone through a similar process in the past (lymph node dissection due to breast cancer) and suggestions of the guidelines will be presented in the mobile application. In arm volume measurement, a wearable technology product to be designed in the form of an arm cuff and strain sensors to be placed on the arm will detect the increase in arm circumference. After Summary With the increase in the incidence of cancer in our country and the world, the number of breast cancer survivors is increasing rapidly due to the development of early diagnosis and treatment methods. One of the main problems in breast cancer survivors is lymphedema. Breast cancer-related lymphedema is a condition that can be treated when detected early, but has a very low success rate when detected in advanced stages. Therefore, the prevention and early detection of breast cancer-associated lymphedema is very important. In this project, it is aimed to prevent breast cancer-related lymphedema with the mobile application to be developed and to detect the volume increase in the arm before clinical findings with an arm volume measurement device that will work with this mobile application. The project consists of two main steps; (a)development of the arm volume measuring device and mobile application (b)evaluation of the effectiveness of the products. Five components will be involved in the development of the mobile application. These components are; (I)exercise, (II)education, (III)coping mechanisms, (IV)arm volume measurement/records, and (V)reminder for exercise, measurement, and follow-ups. Exercise videos will include stretching exercises for the shoulder and arm area as recommended in the guides. The training content will be created in line with the guides and opinions will be taken from an expert panel. In support of coping mechanisms, existing problem areas in people will be determined with a qualitative study. People who have gone through a similar process in the past will be asked about the coping strategies they have developed for these problem areas. Themes obtained from patients who have gone through a similar process in the past (lymph node dissection due to breast cancer) and suggestions of the guidelines will be presented in the mobile application. In arm volume measurement, a wearable technology product to be designed in the form of an arm cuff and strain sensors to be placed on the arm will detect the increase in arm circumference. After measuring the arm circumference with the sensors located every five centimeters, the arm volume will be calculated with the cylindrical volume calculation method. When there is an increase of 5% or more in the arm of the individual (preclinical lymphedema), a notification will be sent to the person and his/her physician via the mobile application. The person will also be able to follow the past measurement results via the mobile application. Evaluation of the efficacy of the product will be based on a pilot randomized controlled trial, a reproducibility study, and patient feedback. This product to be developed will provide a new arm volume measurement method that will reduce patients' hospital admissions and will contribute to the prevention and early detection of lymphedema.

DETAILED DESCRIPTION:
Stage 1 - Development of Arm Volume Measurement Device and Mobile Application; In this stage, the preparation of the mobile application content, the development of the arm volume measurement device and the establishment of the connection unit will be started. Then, these systems will be brought together and feedback will be received from the survivors. In this process, initially 5 lines of work will be carried out simultaneously in the research. These tasks are (1) creation of exercise content and videos, (2) creation of training content, (3) determination of the problem areas experienced by breast cancer survivors through qualitative interviews and determination of the solutions applied by the survivors themselves for these problem areas, (4) development and calibration of the strain sensor and connection unit, 5) expert and user opinions will be taken for the developed mobile application.

Stage 2 - Evaluation of the Effectiveness of the Developed Product; Three simultaneous evaluations will be used in this phase. For this, there will be two research and one end-user feedback. These are; (6) feedback from survivors on satisfaction, usefulness and usefulness after using the product, (7) a pilot randomised controlled trial to evaluate the effectiveness of the developed product and (8) a reproducibility study comparing the developed product with the existing volume measurement method.

ELIGIBILITY:
Inclusion Criteria:

* To agree to take part in the research,
* Breast surgery including lymph node dissection within the last 6 months,
* To be 18 years of age or older,
* To be able to communicate in Turkish,
* Using a smartphone with Android operating system,
* No cognitive/cognitive impairment (electronic records of patients will be taken as basis)

Exclusion Criteria:

* Patients who do not meet the inclusion criteria will be excluded from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who had breast surgery including lymph node dissection within the last 6 months
Enrollment: 14 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Disability of Arm, Shoulder and Hand- DASH | It will be applied to the participants at baseline, as well as at the 25th month and 33th month follow ups.
  The first section contains 30 questions, of which 21 questions assess difficulties experienced in activities of daily living, 5 questions assess symptoms and 4 questions assess social functioning, work, sleep and patient confidence. This section determines the patient's function/symptom status and is referred to as the DASH-FS.
Adult Life Quality Scale in Cancer Survivors | It will be applied to the participants at baseline, as well as at the 25th month and 33th month follow ups.
  Consisting of 47 items and 12 sub-dimensions, the items in the scale are answered in 7-point Likert type. The scale consists of two parts: general and cancer-specific quality of life. Of these 12 sub-dimensions, 7 are related to general quality of life and 5 are related to cancer-specific quality of life.
Positive Affectivity, Negative Affectivity Scale - PANAS | It will be applied to the participants at baseline, as well as at the 25th month and 33th month follow ups.
  The 10 affect states of Excited, Strong, Enthusiastic, Proud, Alert, Inspired, Determined, Active, Concerned, and Attentive measure positive affect; the 10 affect states of Distressed, Unhappy, Guilty, Frightened, Hostile, Irritable, Embarrassed, Nervous, Agitated, and Scared measure negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: İsmail Toyğar, PhD; RN, Principal Investigator — Muğla Sıtkı Koçman University

IPD SHARING:
Plan to Share IPD: Undecided